CLINICAL TRIAL: NCT04172987
Title: Effect of Tirzepatide on Oral Contraceptive Pharmacokinetics in Healthy Female Subjects
Brief Title: A Study of the Effect of Tirzepatide on How the Body Handles Birth Control Pills in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17103; I8F-MC-GPGR (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2022-06

CONDITIONS: Healthy
MeSH Terms: interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ethinyl Estradiol + Norgestimate (EE/NGM) Alone (Period 1) (Experimental): Participants received a 28-day packet of a combination oral contraceptive (OC) containing 21 days of tablets that consist of active ingredients (0.035 mg ethinyl estradiol (EE) and 0.25 mg norgestimate (NGM)) self-administered orally once-daily (QD) on Day 1 to Day 21, and 7 days of non-active tablets self-administer orally QD on Day 22 to Day 28 approximately the same time each day.
  Interventions: Drug: EE/NGM
- EE/NGM + Tirzepatide (Period 2) (Experimental): Participants received a 28-day packet of a combination OC containing 21 days of tablets that consist of active ingredients (0.035 mg EE and 0.25 mg NGM) self-administered orally QD on Day 1 to Day 21, and 7 days of non-active tablets self-administer orally QD on Day 22 to Day 28 approximately the same time each day and a single dose 5 mg tirzepatide administered subcutaneously (SC).
  Interventions: Drug: Tirzepatide; Drug: EE/NGM

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: EE/NGM + Tirzepatide (Period 2)
Drug: EE/NGM — Combination oral contraceptive administered orally

SUMMARY:
The purpose of this study is to look at how the body processes the commonly prescribed birth control pill, ethinylestradiol + norgestimate (EE/NGM), in healthy female participants and the effect of tirzepatide on how EE/NGM is processed by the body. Information about any side effects that may occur will also be collected.

Screening is required within 28 days prior to the start of the study. For each participant, the study will last about 20 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy females as determined by medical history, physical examination, and other screening procedures
* Have a body mass index (BMI) equal to or above 18.5 kilograms per meter squared (kg/m²), at screening
* Are not intending to start a family within 2 months after the study

Exclusion Criteria:

* Have known allergies to either tirzepatide or ethinylestradiol or norgestimate or related compounds
* Have a medical condition or medical history that precludes the taking of combined oral contraceptives
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis), elevation in serum amylase or lipase or gastrointestinal (GI) disorder (eg, relevant esophageal reflux or gall bladder disease) or any GI disease which impacts gastric emptying (eg, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by glucagon-like peptide-1 (GLP-1) analogs or dipeptidyl peptidase IV (DPP-IV) inhibitors
* Have used hormonal implants or received hormonal injections in the past 12 months
* Unwilling to comply with smoking restrictions during the study
* Is a known user of drugs of abuse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Lead In Period and Period 1:
  Participants received a 28-day packet of a combination oral contraceptive (OC) containing 21 days of tablets that consist of active ingredients (0.035 mg ethinyl estradiol (EE) and 0.25 mg norgestimate (NGM)) self-administered orally once-daily (QD) on Day 1 to Day 21, and 7 days of non-active tablets self-administer orally QD on Day 22 to Day 28 approximately the same time each day.
  Period 2:
  Participants received a 28-day packet of a combination OC containing 21 days of tablets that consist of active ingredients (0.035 mg EE and 0.25 mg NGM) self-administered orally QD on Day 1 to Day 21, and 7 days of non-active tablets self-administer orally QD on Day 22 to Day 28 approximately the same time each day and a single dose 5 mg tirzepatide administered subcutaneously (SC).
Period: Lead In Period
Arm/Group | Overall Study
Started | 40
Received at Least One Dose of OC | 40
Completed | 38
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Period: Period 1
Arm/Group | Overall Study
Started | 38
Received at Least One Dose of OC | 38
Completed | 37
Not Completed | 1
Not completed — Physician Decision | 1
Period: Period 2
Arm/Group | Overall Study
Started | 37
Received at Least One Dose of OC | 37
Received at Least 1 Dose of Tirzepatide | 28
Completed | 28
Not Completed | 9
Not completed — Adverse Event | 5
Not completed — Dosing Termination by Sponsor | 4

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of oral contraceptive or tirzepatide.
Groups:
- Overall Study: Lead In Period and Period 1:
  Participants received a 28-day packet of a combination OC containing 21 days of tablets that consist of active ingredients (0.035 mg EE and 0.25 mg NGM) self-administered QD on Day 1 to Day 21, and 7 days of non-active tablets self-administer orally QD on Day 22 to Day 28 approximately the same time each day.
  Period 2:
  Participants received a 28-day packet of a combination OC containing 21 days of tablets that consist of active ingredients (0.035 mg EE and 0.25 mg NGM) self-administered orally QD on Day 1 to Day 21, and 7 days of non-active tablets self-administer orally QD on Day 22 to Day 28 approximately the same time each day and a single dose 5 mg tirzepatide administered SC.
Arm/Group | Overall Study
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 20
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Period 1 and Period 2, Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) Within 1 Dosing Interval (AUC[0-tau]) of Ethinylestradiol (EE)
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) Within 1 Dosing Interval (AUC[0-tau]) of Ethinylestradiol (EE)
Time Frame: Period 1 and Period 2: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48 hours postdose
Population: Period 1 and Period 2: All participants who received at least one dose of oral contraceptive or tirzepatide and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram hour per milliliter (pg*h/mL)
Groups:
- OC (0.035 mg EE and 0.25 mg NGM): Participants received a 28-day packet of a combination OC containing 21 days of tablets that consist of active ingredients (0.035 mg EE and 0.25 mg NGM) self-administered QD on Day 1 to Day 21, and 7 days of non-active tablets self-administer orally QD on Day 22 to Day 28 approximately the same time each day.
- OC (0.035 mg EE and 0.25 mg NGM) + 5 mg Tirzepatide: Participants received a 28-day packet of a combination OC containing 21 days of tablets that consist of active ingredients (0.035 mg EE and 0.25 mg NGM) self-administered orally QD on Day 1 to Day 21, and 7 days of non-active tablets self-administer orally QD on Day 22 to Day 28 approximately the same time each day and a single dose 5 mg tirzepatide administered SC.
Arm/Group | OC (0.035 mg EE and 0.25 mg NGM) | OC (0.035 mg EE and 0.25 mg NGM) + 5 mg Tirzepatide
Number analyzed (Participants) | 35 | 21
picogram hour per milliliter (pg*h/mL) | 966 (40) | 811 (41)

2. Primary Outcome: Period 1 and Period 2, PK: Maximum Concentration (Cmax) of EE
Description: PK: Cmax of EE
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per milliliter pg/mL
Arm/Group | OC (0.035 mg EE and 0.25 mg NGM) | OC (0.035 mg EE and 0.25 mg NGM) + 5 mg Tirzepatide
Number analyzed (Participants) | 35 | 24
picogram per milliliter pg/mL | 119 (33) | 49.6 (63)

3. Primary Outcome: Period 1 and Period 2, PK: Area Under the Concentration Versus Time Curve (AUC) Within 1 Dosing Interval (AUC[0-tau]) of Norelgestromin (NGMN)
Description: PK: Area Under the Concentration Versus Time Curve (AUC) Within 1 Dosing Interval (AUC[0-tau]) of Norelgestromin (NGMN)
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | OC (0.035 mg EE and 0.25 mg NGM) | OC (0.035 mg EE and 0.25 mg NGM) + 5 mg Tirzepatide
Number analyzed (Participants) | 35 | 26
pg*h/mL | 19900 (27) | 14600 (67)

4. Primary Outcome: Period 1 and Period 2, PK: Cmax of Norelgestromin (NGMN)
Description: PK: Cmax of Norelgestromin (NGMN)
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | OC (0.035 mg EE and 0.25 mg NGM) | OC (0.035 mg EE and 0.25 mg NGM) + 5 mg Tirzepatide
Number analyzed (Participants) | 35 | 26
pg/mL | 2070 (27) | 892 (74)

ADVERSE EVENTS:
Time Frame: Lead-In Up To 15 Weeks
Description: All participants who received OC and tirzepatide.
Groups:
- Lead-in: OC ( 0.035 mg EE and 0.25 mg NGM); Period 1: OC ( 0.035 mg EE and 0.25 mg NGM): Participants received a 28-day packet of a combination oral contraceptive (OC) containing 21 days of tablets that consist of active ingredients (0.035 mg ethinyl estradiol (EE) and 0.25 mg norgestimate (NGM)) self-administered orally once-daily (QD) on Day 1 to Day 21, and 7 days of non-active tablets self-administer orally QD on Day 22 to Day 28 approximately the same time each day.
- Period 2: OC ( 0.035 mg EE and 0.25 mg NGM) + 5 mg Tirzepatide: Participants received a 28-day packet of a combination OC containing 21 days of tablets that consist of active ingredients (0.035 mg EE and 0.25 mg NGM) self-administered orally QD on Day 1 to Day 21, and 7 days of non-active tablets self-administer orally QD on Day 22 to Day 28 approximately the same time each day and a single dose 5 mg tirzepatide administered SC.
Arm/Group | Lead-in: OC ( 0.035 mg EE and 0.25 mg NGM) | Period 1: OC ( 0.035 mg EE and 0.25 mg NGM) | Period 2: OC ( 0.035 mg EE and 0.25 mg NGM) + 5 mg Tirzepatide
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/38 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38 | 0/28
Other Adverse Events (participants affected / at risk) | 9/40 | 10/38 | 18/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-in: OC ( 0.035 mg EE and 0.25 mg NGM) (N=40) | Period 1: OC ( 0.035 mg EE and 0.25 mg NGM) (N=38) | Period 2: OC ( 0.035 mg EE and 0.25 mg NGM) + 5 mg Tirzepatide (N=28)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (5)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (2) | 11 (13)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (6)
Chills (General disorders) | 0 (0) | 0 (0) | 3 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 3 (3)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 4 (5) | 5 (5)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 2 (3) | 1 (1) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT04172987/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/87/NCT04172987/SAP_001.pdf